CLINICAL TRIAL: NCT04355663
Title: Neuroproprioceptive Facilitation and Inhibition Physical Therapy Activates Adaptive and Plastic Changes in the Central Nervous System
Brief Title: Neuroproprioceptive "Facilitation, Inhibition" and Brain Plasticity
Acronym: NEFAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, assoc. prof. Kamila Řasová, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VP/22/0/2014
Record Dates: First submitted 2020-04-18; First posted 2020-04-21 (Actual); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; physical therapy; white matter integrity; neuroproprioceptive "facilitation, inhibition"; functional recovery; network reorganization; neurohormones; dehydroepiandrosterone
MeSH Terms: conditions — Multiple Sclerosis; Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor program activating therapy (Experimental): MPAT is method developed and verified by our team. In this therapy, patients are corrected into a postural position where the joints are functionally centered. Somatosensory (manual and verbal) stimuli are then applied to activate motor programs in the brain, which then lead to the co-contraction of the patient's whole body when laying, sitting, standing up or moving forward. Activated programs are repeated under various conditions and in different situations and environments to teach the patients to automatically use the acquired motor skills in daily life. Therapy was realized within the ambulatory area of the Department of Neurology at Kralovske Vinohrady University Hospital in Prague.
  Interventions: Behavioral: Motor program activating therapy
- Vojta's reflex locomotion (Experimental): VRL is a standard approach for patients with MS in the Czech Republic. In the therapy, global patterns of the reflex locomotion are activated by stimulation of specific zones, with the individual placed in a precisely determined initial position (supine, prone and side laying, low kneeling position). These movement patterns have the qualities of the forward movement (locomotion) and the movement responses are precisely defined. Reflex locomotion (reflex turning and reflex creeping) is used in therapy to activate involuntarily responses of muscle function, which are necessary for spontaneous movements. Therapy was realized at the Department of Rehabilitation and Sport Medicine at Motol University Hospital.
  Interventions: Behavioral: Vojta's reflex locomotion
- Functional electric stimulation (Experimental): Functional electric stimulation in the postural corrected position was developed at our workplace. Participants first underwent individual two-hour session consisting of postural correction using MPAT and the device (The WalkAide® System, Innovative Neurotronics Inc., 4999 Aircenter Circle, Suite 103 Reno, NV 89502, USA) programming (28). Patients received the device to use as much as they felt they were able to during their normal daily living activities thereafter.
  Interventions: Behavioral: Functional electric stimulation

INTERVENTIONS:
Behavioral: Motor program activating therapy — Pacients underwent two months' therapy consisted of 16 face-to-face sessions (1 hour, twice a week for two months).
  Arms: Motor program activating therapy
Behavioral: Vojta's reflex locomotion — Pacients underwent two months' therapy consisted of 16 face-to-face sessions (1 hour, twice a week for two months).
  Arms: Vojta's reflex locomotion
Behavioral: Functional electric stimulation — Pacients uderwent two months' therapy. They used the whole time Functional electric stimulation during activities of daily living and underwent 2 individual sessions of Motor program activating therapy.
  Arms: Functional electric stimulation

SUMMARY:
This study investigates whether neuroproprioceptive "facilitation, inhibition" physical therapy induces plastic and adaptive processes of the CNS (white matter integrity changes), if they relate to clinical improvement, and whether therapeutic effect differs between different kinds of therapies.

DETAILED DESCRIPTION:
In the Multi-Arm Parallel-Group Exploratory Trial, patients with multiple sclerosis were divided into three groups by an independent study coordinator, and underwent three kinds of neuroproprioceptive "facilitation, inhibition" physical therapy. At baseline and after the end of the two months' therapeutic program, a blinded assessor evaluated clinical outcomes and data from DTI .

ELIGIBILITY:
Inclusion Criteria:

* prevailed spastic paraparesis, stable clinical status and treatment in the preceding 3 months determined by neurologist,
* Expanded Disability Status Scale score (EDSS) max. 7.5

Exclusion Criteria:

* other neurological disease or conditions disabling movement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Řasová, Ph.D., Principal Investigator — Third Faculty of Mecicine, Charles Univerzity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasova K, Buckova B, Prokopiusova T, Prochazkova M, Angel G, Markova M, Hruskova N, Stetkarova I, Spanhelova S, Mares J, Tintera J, Zach P, Musil V, Hlinka J. A Three-Arm Parallel-group Exploratory Trial documents balance improvement without much evidence of white matter integrity changes in people with multiple sclerosis following two months ambulatory neuroproprioceptive "facilitation and inhibition" physical therapy. Eur J Phys Rehabil Med. 2021 Dec;57(6):889-899. doi: 10.23736/S1973-9087.21.06701-0. Epub 2021 Feb 10. PMID 33565742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was realized between May 2015 and May 2017 at Department of Neurology, Facuty Hospital Royal Vineyard. MS patients were divided into three groups by an independent study coordinator according to availability of each therapist (in Groups 1 and 2) and amount of FES devices to borrow (in Group 3), and underwent three kinds of PT.
Pre-assignment Details: 120 people were initially assessed for eligibility. 24 people did not fit to inclusion criteria, 1 did decline to participate and 1 injured. 92 were allocated into three groups.
Groups:
- Motor Program Activating Therapy: MPAT is method developed and verified by our team. In this therapy, patients are corrected into a postural position where the joints are functionally centered. Somatosensory (manual and verbal) stimuli are then applied to activate motor programs in the brain, which then lead to the co-contraction of the patient's whole body when laying, sitting, standing up or moving forward.
  16 face-to-face sessions (1 hour, twice a week for two months). Group 3 used the whole time Functional electric stimulation during activities of daily living and underwent 2 individual sessions.
- Vojta's Reflex Locomotion: VRL is a standard approach for patients with MS in the Czech Republic. In the therapy, global patterns of the reflex locomotion are activated by stimulation of specific zones, with the individual placed in a precisely determined initial position (supine, prone and side laying, low kneeling position).
  16 face-to-face sessions (1 hour, twice a week for two months). Group 3 used the whole time Functional electric stimulation during activities of daily living and underwent 2 individual sessions.
- Functional Electric Stimulation: Functional electric stimulation in the postural corrected position was developed at our workplace. Participants first underwent individual two-hour session consisting of postural correction using MPAT and the device (The WalkAide® System, Innovative Neurotronics Inc., 4999 Aircenter Circle, Suite 103 Reno, NV 89502, USA) programming (28). Patients received the device to use as much as they felt they were able to during their normal daily living activities thereafter.
  Patients used the whole time Functional electric stimulation during activities of daily living and underwent 2 individual sessions.
Period: Overall Study
Arm/Group | Motor Program Activating Therapy | Vojta's Reflex Locomotion | Functional Electric Stimulation
Started | 42 | 29 | 21
Completed | 40 | 14 | 17
Not Completed | 2 | 15 | 4
Not completed — Physician Decision | 2 | 7 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 8 | 3

BASELINE CHARACTERISTICS:
Population: 92 patients were allocated into three groups; from these 71 participants finished their therapeutic programs. Data of ten patients were discarded upon the visual control, due to the low quality of DTI acquisition resulting in 61 participants entering the central analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Motor Program Activating Therapy | Vojta's Reflex Locomotion | Functional Electric Stimulation | Total
Number analyzed (Participants) | 42 | 29 | 21 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 29 | 21 | 92
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10.7) | 42.3 (10.5) | 46.15 (10.1) | 48.11 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 19 | 12 | 61
  Male | 12 | 10 | 9 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 29 | 21 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 35 | 13 | 13 | 61
length of disease [Mean (Standard Deviation); unit: years] | 14.2 (7.4) | 8.38 (5.1) | 13.15 (6.1) | 12.72 (7.0)
EDSS [Median (Inter-Quartile Range); unit: units on a scale] — The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability (minimum 0 - the worse, maximum 10 - the best). Scoring is based on an examination by a neurologist.
  units on a scale | 4 [1 to 7] | 4 [1 to 6] | 4 [2 to 7] | 4 [1 to 7]

OUTCOME MEASURES:

1. Primary Outcome: White Matter Integrity
Description: Magnetic resonance imaging on a 3T magnetic resonance scanner (Siemens Trio Tim, Erlangen, Germany) using a 12-channel phased-array head coil. A diffusion tensor was fitted to each voxel of the brain, and a fractional anisotropy (FA) map was created for each subject. The images were further analyzed using tract-based spatial statistics (TBSS).
  Fractional anisotropy (FA) is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions. FA is a measure often used in diffusion imaging where it is thought to reflect fiber density, axonal diameter, and myelination in white matter. The FA is an extension of the concept of eccentricity of conic sections in 3 dimensions, normalized to the unit range.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Program Activating Therapy | Vojta's Reflex Locomotion | Functional Electric Stimulation
Number analyzed (Participants) | 42 | 29 | 21
score on a scale | 0.5023 (0.0293) | 0.5168 (0.0266) | 0.4747 (0.0293)

2. Secondary Outcome: Berg Balance Scale, BBS
Description: 14 items objective measure of static balance and risk of falls (0 the best, 56 the worse)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Program Activating Therapy | Vojta's Reflex Locomotion | Functional Electric Stimulation
Number analyzed (Participants) | 42 | 29 | 21
score on a scale | 49.79 (8.1) | 47.92 (9.8) | 32.76 (11.2)

3. Secondary Outcome: Timed up and go Test, TUG
Description: time necessary to stand up, go 3 meters, turn around, go back and sit to chair (longer time in seconds is worse function)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Motor Program Activating Therapy | Vojta's Reflex Locomotion | Functional Electric Stimulation
Number analyzed (Participants) | 42 | 29 | 21
sec | 10.15 (5.8) | 10.31 (5.6) | 16.88 (10.8)

4. Secondary Outcome: the 12-item Multiple Sclerosis Walking Scale, MSWS - 12
Description: The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
  A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Program Activating Therapy | Vojta's Reflex Locomotion | Functional Electric Stimulation
Number analyzed (Participants) | 42 | 29 | 21
score on a scale | 61.57 (12.7) | 59.77 (18.4) | 73.94 (20.2)

5. Secondary Outcome: the 29-item Multiple Sclerosis Impact Scale, MSIS -29
Description: a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motor Program Activating Therapy | Vojta's Reflex Locomotion | Functional Electric Stimulation
Number analyzed (Participants) | 42 | 29 | 21
score on a scale | 32.93 (8.7) | 33.38 (13.3) | 43.47 (12.6)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 2 months
Arm/Group | Vojta's Reflex Locomotion | Motor Program Activating Therapy | Functional Electric Stimulation
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/42 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/42 | 1/21
Other Adverse Events (participants affected / at risk) | 0/29 | 0/42 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vojta's Reflex Locomotion (N=29) | Motor Program Activating Therapy (N=42) | Functional Electric Stimulation (N=21)
falling (Nervous system disorders) | 0 | 0 | 1 — an increased number of falls

LIMITATIONS AND CAVEATS:
Different availability to undergo therapy and limited supply of the FES device leading to non-uniform distribution of participants within groups; Technical problems with measurement of DTI leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT04355663/Prot_SAP_000.pdf